CLINICAL TRIAL: NCT00894049
Title: A Multicenter Prospective Randomized Study Comparing Non Myeloablative (Flu-TBI) and Reduced Intensity (FLU-BU-ATG) Conditioning in Allogenic Transplantation
Brief Title: A Study Comparing Non Myeloablative (Flu-TBI) and Reduced Intensity (FLU-BU-ATG) Conditioning in Allogenic Transplantation
Acronym: ITAC02-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITAC02-01
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Allograft; Allogeneic Cell Transplantaion; Hematological Malignancy; Solid Tumor
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flu-Bu-ATG (Experimental): Fludarabine (30mg/m²/5 days) Oral Busulfan (8 mg/kg over 2 days) Thymoglobuline (2.5 mg/m²/1day).
  Interventions: Drug: reduced intensity conditionings
- Fluda-TBI (Experimental): Fludarabine (25mg/m²/ 3 days) 2 Gy TBI
  Interventions: Drug: reduced intensity conditionings

INTERVENTIONS:
Drug: reduced intensity conditionings — comparison of non myeloablative (Flu-TBI) and reduced intensity (FLU-BU-ATG)

SUMMARY:
This study is a prospective comparison between 2 popular regimens based on reduced intensity or non-myeloablative approaches to define the optimal myeloablative and/or immu-nonsuppressive association for reduced intensity conditionings (RIC).

Flu-Bu-ATG (Study A) associated Fludarabine (30mg/m²/5 days), Oral Busulfan (8 mg/kg over 2 days) and Thymoglobuline (2.5 mg/m²/1day).

Flu-TBI (Study B) consisted of Fludarabine (25mg/m²/ 3 days) and 2 Gy total body irradiation (TBI).

A randomization of 2 phase study according to the methodology developed by Liu et al (Liu, 1993 and 2001) for the evaluation of multiple innovative approaches.

Primary endpoint is one year overall survival (OS). Stopping rules included excessive engraftment failure and trans-plant related mortality ratio. Data are yearly reviewed by an independent safety review board (ISRB).

Inclusion criteria are patients presenting a hematological malignancy, eligible for non myeloablative allo stem cell transplantation (SCT), aged between 18 and 65, with a suitable HLA identical sibling. All patients and donors are included after giving written informed consent.

Protocol was submitted and accepted by the ethical committee and the AFFSSAPS cellular therapies committee (national agency).

ELIGIBILITY:
Inclusion Criteria:

* hematological malignancy or solid tumor,
* eligible for non myeloablative allogenic transplantation,
* aged between 18 and 65,
* with a suitable HLA identical sibling

Exclusion Criteria:

* contra-indication to allogenic transplantation
* pregnant women or breast feeding
* active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2002-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
one year overall survival (OS) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Didier BLAISE, PUPH, Principal Investigator — Institut Paoli-Calmettes
Locations (5):
- France (5):
  - CHU, Bordeaux Pessac
  - CHU, Clermont-Ferrand
  - CHU, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU, Montpellier

REFERENCES:
- See also: official site of the sponsor — http://www.institutpaolicalmettes.fr/